CLINICAL TRIAL: NCT00966615
Title: The Effect of Neutral Peritoneal Dialysis Solution With Minimal Glucose-Degradation-Product on the Fluid Status and Body Composition - A Randomized Control Trial
Brief Title: The Effect of Neutral Peritoneal Dialysis (PD) Solution With Minimal Glucose-Degradation-Product (GDP) on Fluid Status and Body Composition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Balance BCM
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Renal Failure; ESRD; Cardiovascular Disease
Keywords: malnutrition; fluid status; survival
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Cardiovascular Diseases; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance group (Experimental): peritoneal dialysis with neutral peritoneal dialysis solution with minimal glucose-degradation-product
  Interventions: Other: double-chamber bag Stay-Safe Balance system
- Control group (Active Comparator): conventional PD solution
  Interventions: Other: glucose-based dialysis solution

INTERVENTIONS:
Other: double-chamber bag Stay-Safe Balance system — 2-L exchange; three times a day
  Other Names: Stay-Safe Balance system
  Arms: Balance group
Other: glucose-based dialysis solution — 2-L exchange; three times a day
  Other Names: Stay-Safe, Fresenius
  Arms: Control group

SUMMARY:
Chronic utilization of bio-incompatible peritoneal dialysis (PD) solution has been implicated as a cause of progressive loss of peritoneal permeability and recurrent fluid overload in PD patients. Previous studies show that PD solution with neutral pH and low GDP resulted in a superior profile of PD effluent mesothelial cell marker and a lower degree of systemic inflammation as compared to conventional PD solution. The investigators propose a prospective randomized control study to compare the arterial stiffness, nutrition and body fluid status between PD patients treated with conventional solution and those with neutral pH low GDP solution. The investigators plan to study 100 new PD patients. They will be randomized to be treated with neutral pH low GDP solution or conventional solution. All patients will be followed for 52 weeks. In addition to routine clinical measurements, the investigators will measure their body water composition by bioimpedance spectroscopic method, arterial pulse wave velocity by pressure transduction method, as well as radiographic parameters of intravascular volume status, based on the routine chest radiograph. The study would help to define the clinical benefit of biocompatible PD solution.

DETAILED DESCRIPTION:
(see above)

ELIGIBILITY:
Inclusion Criteria:

* new adult continuous ambulatory peritoneal dialysis (CAPD) patients, both diabetic and non-diabetic

Exclusion Criteria:

* unlikely to survive, planned to have elective living-related kidney transplant, or transfer to other renal center within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
body composition | 52 weeks
arterial pulse wave velocity | 52 weeks

SECONDARY OUTCOMES:
nutritional and adequacy indices | 52 weeks
peritoneal transport characteristics | 52 weeks
residual renal function | 52 weeks
peritonitis-free survival, actuarial and technique survival | 52 weeks
hospitalization | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong; Philip KT Li, MD, Study Director — Prince of Wales Hospital, Shatin, Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Derived] Szeto CC, Kwan BC, Chow KM, Cheng PM, Kwong VW, Choy AS, Law MC, Leung CB, Li PK. The Effect of Neutral Peritoneal Dialysis Solution with Low Glucose-Degradation-Product on the Fluid Status and Body Composition--A Randomized Control Trial. PLoS One. 2015 Oct 28;10(10):e0141425. doi: 10.1371/journal.pone.0141425. eCollection 2015. PMID 26510186